CLINICAL TRIAL: NCT07349472
Title: Clinical Study Evaluating Safety and Efficacy of Pentoxifylline in Patients With Ulcerative Colitis
Brief Title: Pentoxifylline in Patients With Ulcerative Colitis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ihab Elsayed Hassan (Other)
Responsible Party: Sponsor-Investigator, Ihab Elsayed Hassan, Lecturer, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 87459
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Mesalamine; Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Group 1 (Placebo Group): Participants in this arm were administered an inert placebo capsule twice per day, in combination with mesalamine at a total daily dose of 3 g, given as 1 g three times daily
  Interventions: Drug: Mesalamine
- Pentoxifylline group (Active Comparator): Group 2 (PTX Group): Individuals assigned to this group received PTX at a dose of 400 mg twice daily, together with mesalamine 1 g taken three times daily.
  Interventions: Drug: Mesalamine; Drug: Pentoxifylline

INTERVENTIONS:
Drug: Mesalamine — Mesalamine is the standard first line treatment of ulcerative colitis
Drug: Pentoxifylline — Pentoxifylline (PTX), a methylxanthine derivative and non-selective phosphodiesterase inhibitor, has been extensively studied for its anti-inflammatory and immunomodulatory actions. It inhibits TNF-α production at the transcriptional level and downregulates several inflammatory cytokines, including IL-1β, IL-6, and interferon-γ
  Arms: Pentoxifylline group

SUMMARY:
Ulcerative colitis (UC) is a persistent, idiopathic form of inflammatory bowel disease (IBD) marked by uninterrupted inflammation of the colon's mucosal lining, usually starting at the rectum and progressing proximally in a continuous manner. It manifests clinically with recurrent episodes of abdominal pain, bloody diarrhea, urgency, tenesmus, and weight loss. The precise cause of UC is still unknown; however, it is thought to arise from a multifactorial interaction involving genetic susceptibility, immune system dysregulation, disturbances in gut microbiota composition, and various environmental factors.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Both male and female will be included
* Negative pregnancy test and effective contraception.
* Mild and moderate UC patients

Exclusion Criteria:

* Breast feeding
* Significant liver and kidney function abnormalities
* Diabetic patients
* Colorectal cancer patients
* Patients with severe UC
* Patients taking rectal or systemic steroids
* Patients taking immunosuppressives or biological therapies
* Addiction to alcohol and / or drugs
* Known allergy to the studied medications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2027-01-20 (Estimated); Study Completion 2027-02-20 (Estimated)

PRIMARY OUTCOMES:
Change in partial Mayo score | 6 months
  The Partial Mayo Score (PMS) was utilized to evaluate disease activity in patients with UC. This non-invasive index comprises three components: stool frequency, rectal bleeding, and the physician's global assessment, yielding a total score between 0 and 9

SECONDARY OUTCOMES:
Change in inflammatory bowel disease questionnaire-32 (IBDQ-32) | 6 months
  The IBDQ-32 is the most widely used tool for evaluating disease-specific quality of life in randomized clinical trials involving UC. It measures four domains: emotional function, social function, bowel symptoms, and systemic symptoms
Change in level of fecal calprotectin | 6 months
  Fecal calprotectin is a non-invasive marker used as a prognostic tool in colitis

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University, Al Fayyum, Egypt